CLINICAL TRIAL: NCT02594735
Title: Abatacept for the Treatment of Refractory Juvenile Dermatomyositis
Brief Title: Abatacept in Juvenile Dermatomyositis
Acronym: AID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Rodolfo Curiel, Dr. Rodolfo V. Curiel, MD, Associate Professor of Medicine, Division of Rheumatology; Director, Myositis Center, George Washington University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 111418
Record Dates: First submitted 2015-10-21; First posted 2015-11-03 (Estimated); Results first posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Dermatomyositis
Keywords: Juvenile dermatomyositis; inflammatory myopathies; Orencia; Abatacept
MeSH Terms: conditions — Dermatomyositis; Myositis | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label (One Arm) (Other): A patient's participation in this study will last approximately 24 weeks ( screening visit and 5 intervention visits) with possible extension to 48 weeks. At screening, participants will have a physical exam, muscle strength assessment, blood and urine collection, and chest x-ray; they will also be asked to complete several questionnaires. All participants will receive each week subcutaneous injection of Abatacept. During intervention phase of the trial, muscle strength testing, physical exam, disease activity measurements, blood and urine collection, and muscle MRI will be performed. Participants will also be asked to complete several questionnaires. Participants will be also monitored closely for for serious drug related side effects.
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — Study participation will consist of a screening visit and 5 protocol visits over six months (week 0, week 6, week 12, week 18, and week 24) for each subject, and phone follow-up (week 2, week 4, week 8, week 10, week 14, week 16, week 20, and week 22). At Visit 1, which will be treatment initiation, eligible subjects will be instructed on the use and side effects of subcutaneous abatacept and will be started on the study drug (abatacept 125 mg SQ weekly for subjects with body weight ≥ 50 KG or abatacept 87.5mg SQ for subjects with body weight < 50 KG).
  Other Names: Orencia

SUMMARY:
The purpose of this study is to assess the safety and efficacy of subcutaneous abatacept in 10 patients seven years of age and older with refractory JDM.

DETAILED DESCRIPTION:
JDM is a chronic systemic autoimmune disease with a predominance of muscle and skin inflammation of unknown etiology and varying prognosis. Children with JDM unresponsive to corticosteroids or other immunosuppressive medications face poor clinical and functional outcome and suffer various sequelae of the disease. Abatacept is a fully human soluble recombinant protein consisting of the cytotoxic T cell Lymphocyte Antigen-4 (CTLA4) fused with Fc region of human IgG1 that has been modified to prevent complement fixation and antibody-dependent cellular cytotoxicity. Abatacept binds specifically to the CD80 (B7-1) and CD86 (B7-2) molecules, those expressed on antigen-presenting cells (APCs). Upon engagement of CTLA4 to CD80 or CD86, the resultant inhibition of signal transduction inhibits T cell activation.. The rationale for use of Abatacept in the therapy of JDM includes the expression of CTLA4, CD28, CD86, and CD40 on inflammatory cells of muscle biopsies of patients with DM, as well as CTLA4 and CD28 on muscle cells.

A patient's participation in this study will last approximately 24 weeks with possible extension to 48 weeks. At screening, participants will have a physical exam, muscle strength assessment, blood and urine collection, and chest x-ray; they will also be asked to complete several questionnaires. All participants will receive each week subcutaneous injection of Abatacept. Each injection will be given on an outpatient basis.

There will be a total of 6 study visits. All participants will visit the outpatient clinic at selected time points for muscle strength testing, a physical exam, disease activity measurements, blood and urine collection, and muscle MRI; they will also be asked to complete several questionnaires. During the study, participants will be monitored closely for improvement or worsening of their disease and for serious drug related side effects.

Eligibility Ages Eligible for Study: ≥ 7 years and older Genders Eligible for Study: Both Race/Ethnic Backgrounds Eligibility for Study: No restrictions

ELIGIBILITY:
Inclusion Criteria:

1. Adults with definite or probable JDM and pediatric patients 7 years of age and older with definite or probable JDM.
2. Body weight of at least 25 kg (or at least 55 lbs) and age ≥ 7 years of age.
3. Patients must reside within the United States or Canada.
4. Refractory myositis, as defined by the intolerance to or an inadequate response to corticosteroids plus an adequate regimen of at least one other immunosuppressive agent, including azathioprine, methotrexate, IVIG, mycophenolate mofetil, cyclophosphamide, tacrolimus or cyclosporine A, or a biologic therapy. The definition of intolerance is: side effects that require discontinuation of the medication or an underlying condition that precludes the further use of the medication.
5. At least moderately active disease as documented by:

   * MD global VAS with a minimum value of 2.5 cm on a 10 cm scale AND
   * At least 2 other abnormal core set measures listed below:
6. Therapy with prednisone or another glucocorticoid is required, unless there is documented intolerance in the medical record or a medical condition that contraindicates further use of prednisone. The prednisone dose must be stable for at least 4 weeks prior to the screening visit.
7. Background therapy with at least 1 non-corticosteroid immunosuppressive agent is required at a stable dose for at least 6 weeks prior to the screening visit unless there is documentation that the patient is intolerant, which is defined as side effects that require discontinuation of the medication(s) or an underlying condition that precludes the further use of the IS medication.
8. If an immunosuppressive agent was discontinued prior to the screening visit then there must be a:

   * 4 week washout for prednisone or methotrexate
   * 8 week washout for any other IS agent
   * For discontinuation of biologic therapies, a washout of 5 terminal half lives
9. If on hydroxychloroquine or colchicine, the dose should be stable for 6 weeks prior to Visit 1.
10. If on statin or fibric acid derivative agents, the dose should be stable for 6 weeks prior to Visit 1.
11. Ability of patient or parent to complete self-report questionnaires.
12. Men and women of reproductive potential must agree to use a reliable method of birth control during the 24 week duration of the trial described in the reproductive risks section of this protocol (section 4.3). They must also agree to use a reliable method of birth control for 100 days after the last dose of study drug is administered.
13. Patients must agree to forgo immunization with a live vaccine during the course of the study or within 3 months after discontinuation.
14. Patients must have a letter from the referring rheumatologist or specialist supervising the care of the JDM, agreeing to the patient's participation in the study and to continuing to provide care for the patient, including emergency care during the trial.

Core Set Measures:

* An MMT-8 score that is no greater than 125/150
* Patient/Parent Global VAS with a minimum value of 2.0 cm on a 10cm scale
* CHAQ/HAQ disability index with a minimum value of 0.25
* Elevation of at least one of the muscle enzymes [which includes creatine kinase (CK), aldolase, lactate dehydrogenase (LDH), alanine aminotransferase (ALT) and aspartate aminotransferase (AST)] at a minimum level of 1.3 x the upper limit of normal.
* Global extra-muscular disease activity score with a minimum value of 2.0 cm on a 10 cm VAS scale

Exclusion Criteria:

1. Drug-induced myositis (myositis in patients taking medications known to induce myositis-like syndromes, including, but not limited to, statin agents, fibric acid derivatives, and colchicine).
2. Juvenile polymyositis; inclusion body myositis; cancer-associated myositis, defined as the diagnosis of myositis within 2 years of the diagnosis of cancer except basal or squamous cell skin cancer or carcinoma in situ of the cervix if at least 5 years since excision
3. Myositis in overlap with another connective tissue disease (CTD) that precludes the accurate assessment of a treatment response (for example, difficulty in assessing muscle strength in a scleroderma patient with associated myositis)
4. History of receiving a live vaccine 4 weeks prior to initiation of study treatment
5. Joint disease, severe calcinosis, or other musculoskeletal condition, which precludes the ability to quantitate muscle strength.
6. Wheelchair bound patients.
7. Known hypersensitivity to abatacept or prior receipt of abatacept
8. Concomitant illness that would prevent adequate patient assessment or in the investigators opinion pose an added risk for study participants:
9. Recurrent or chronic infections, including HIV, tuberculosis, hepatitis B and C, or TB infection, including contact with a household contact with active tuberculosis (TB) and who did not receive appropriate and documented prophylaxis for TB. (a documented negative Hepatitis B surface antigen and Hepatitis C antibody completed at the screening visit or within 6 weeks prior to screening visit is required)
10. Have had symptomatic herpes zoster or herpes simplex infection (not including simple oral HSV lesions) within 12 weeks prior to entry or during screening period
11. Have a history of disseminated/complicated herpes zoster (for example, multi-dermatomal involvement, ophthalmic zoster, central nervous system (CNS) involvement, post-herpetic neuralgia)
12. Known liver disease (i.e. cirrhosis or other conditions compromising the synthetic function of the liver)
13. Disorders that would preclude accurate assessment of neuromuscular function
14. Cardiomyopathy or arrhythmias that in the investigators opinion poses an additional risk for study participants
15. New York Heart Association Classification III or IV for congestive heart failure
16. Psychiatric illness that precludes compliance or neuromuscular assessment
17. Serum creatinine > 2.0mg/dl
18. Pregnant females or nursing mothers
19. Life threatening illness that would interfere with the patient's ability to complete the study.
20. Known or suspected history of drug or alcohol abuse within the past 6 months as determined by the medical record or patient interview
21. Anticipated poor compliance
22. Participation in another clinical experimental therapeutic study within 30 days of screening visit.
23. Any history or evidence of severe illness or any other condition that would make the patient, in the opinion of the investigator unsuitable for the study.
24. Low total WBC <2.000, platelets < 100,000/mm3; hemoglobin <10 gm/dl
25. History of recurrent infection including active skin infections with calcinosis
26. Subjects with a history of cancer in the last 5 years
27. Subjects who have at any time received treatment with any investigational drug within 28 days (or less than 5 terminal half-lives of elimination) of the day 1 dose of study drug, including waiting until CD19 returns to a detectable level and IgG level is within normal limits (normal serum levels of IgG per reference lab: 7-9 years ≥572 mg/dl, 10-11 yrs ≥698 mg/dl, 12-13 yrs ≥759 mg/dl, 14-15 yrs ≥716 mg/dl,16-19 yrs ≥549 mg/dl, >19 yrs ≥700 mg/dl) for those patients who have received rituximab
28. Concomitant treatment with anti-TNF therapies, rituximab or anakinra or other biologic therapies.
29. Initiation of colchicine and hydroxychloroquine as new drugs during study participation is not allowed.
30. Initiation of statins or fibric acid derivatives during study participation is not allowed.
31. Initiation of an exercise program within 4 weeks of the screening visit. Only a stretching program may be initiated during the study (See section 5.4 Other Restrictions)
32. Prisoners or subjects who are involuntarily incarcerated.
33. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11; Primary Completion 2021-07-16 (Actual); Study Completion 2021-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo V Curiel, MD, Principal Investigator — The George Washington University
Locations (1):
- 2300 M Street, 9th floor. Medical Faculty Associates, The George Washington University., Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Feldman BM, Rider LG, Reed AM, Pachman LM. Juvenile dermatomyositis and other idiopathic inflammatory myopathies of childhood. Lancet. 2008 Jun 28;371(9631):2201-12. doi: 10.1016/S0140-6736(08)60955-1. PMID 18586175
- [Background] Wedderburn LR, Rider LG. Juvenile dermatomyositis: new developments in pathogenesis, assessment and treatment. Best Pract Res Clin Rheumatol. 2009 Oct;23(5):665-78. doi: 10.1016/j.berh.2009.07.007. PMID 19853831
- [Background] Oddis CV, Reed AM, Aggarwal R, Rider LG, Ascherman DP, Levesque MC, Barohn RJ, Feldman BM, Harris-Love MO, Koontz DC, Fertig N, Kelley SS, Pryber SL, Miller FW, Rockette HE; RIM Study Group. Rituximab in the treatment of refractory adult and juvenile dermatomyositis and adult polymyositis: a randomized, placebo-phase trial. Arthritis Rheum. 2013 Feb;65(2):314-24. doi: 10.1002/art.37754. PMID 23124935
- [Background] Nagaraju K, Raben N, Villalba ML, Danning C, Loeffler LA, Lee E, Tresser N, Abati A, Fetsch P, Plotz PH. Costimulatory markers in muscle of patients with idiopathic inflammatory myopathies and in cultured muscle cells. Clin Immunol. 1999 Aug;92(2):161-9. doi: 10.1006/clim.1999.4743. PMID 10444360
- [Background] Murata K, Dalakas MC. Expression of the costimulatory molecule BB-1, the ligands CTLA-4 and CD28, and their mRNA in inflammatory myopathies. Am J Pathol. 1999 Aug;155(2):453-60. doi: 10.1016/s0002-9440(10)65141-3. PMID 10433938
- [Background] Behrens L, Kerschensteiner M, Misgeld T, Goebels N, Wekerle H, Hohlfeld R. Human muscle cells express a functional costimulatory molecule distinct from B7.1 (CD80) and B7.2 (CD86) in vitro and in inflammatory lesions. J Immunol. 1998 Dec 1;161(11):5943-51. PMID 9834075
- [Background] Azuma M, Ito D, Yagita H, Okumura K, Phillips JH, Lanier LL, Somoza C. B70 antigen is a second ligand for CTLA-4 and CD28. Nature. 1993 Nov 4;366(6450):76-9. doi: 10.1038/366076a0. PMID 7694153
- [Background] Schiff M. Subcutaneous abatacept for the treatment of rheumatoid arthritis. Rheumatology (Oxford). 2013 Jun;52(6):986-97. doi: 10.1093/rheumatology/ket018. Epub 2013 Mar 5. PMID 23463804
- [Background] Arabshahi B, Silverman RA, Jones OY, Rider LG. Abatacept and sodium thiosulfate for treatment of recalcitrant juvenile dermatomyositis complicated by ulceration and calcinosis. J Pediatr. 2012 Mar;160(3):520-2. doi: 10.1016/j.jpeds.2011.11.057. Epub 2012 Jan 13. PMID 22244459
- [Background] Musuruana JL, Cavallasca JA. Abatacept for treatment of refractory polymyositis. Joint Bone Spine. 2011 Jul;78(4):431-2. doi: 10.1016/j.jbspin.2011.03.022. Epub 2011 May 7. No abstract available. PMID 21550833
- [Background] Maeshima K, Kiyonaga Y, Imada C, Iwakura M, Hamasaki H, Haranaka M, Ishii K. Successful treatment of refractory anti-signal recognition particle myopathy using abatacept. Rheumatology (Oxford). 2014 Feb;53(2):379-80. doi: 10.1093/rheumatology/ket251. Epub 2013 Aug 6. No abstract available. PMID 23920268
- [Background] Ruperto N, Lovell DJ, Li T, Sztajnbok F, Goldenstein-Schainberg C, Scheinberg M, Penades IC, Fischbach M, Alcala JO, Hashkes PJ, Hom C, Jung L, Lepore L, Oliveira S, Wallace C, Alessio M, Quartier P, Cortis E, Eberhard A, Simonini G, Lemelle I, Chalom EC, Sigal LH, Block A, Covucci A, Nys M, Martini A, Giannini EH; Paediatric Rheumatology International Trials Organisation (PRINTO); Pediatric Rheumatology Collaborative Study Group (PRCSG). Abatacept improves health-related quality of life, pain, sleep quality, and daily participation in subjects with juvenile idiopathic arthritis. Arthritis Care Res (Hoboken). 2010 Nov;62(11):1542-51. doi: 10.1002/acr.20283. Epub 2010 Jul 1. PMID 20597110
- [Background] Rider LG, Giannini EH, Brunner HI, Ruperto N, James-Newton L, Reed AM, Lachenbruch PA, Miller FW; International Myositis Assessment and Clinical Studies Group. International consensus on preliminary definitions of improvement in adult and juvenile myositis. Arthritis Rheum. 2004 Jul;50(7):2281-90. doi: 10.1002/art.20349. PMID 15248228
- [Background] Ruperto N, Pistorio A, Ravelli A, Rider LG, Pilkington C, Oliveira S, Wulffraat N, Espada G, Garay S, Cuttica R, Hofer M, Quartier P, Melo-Gomes J, Reed AM, Wierzbowska M, Feldman BM, Harjacek M, Huppertz HI, Nielsen S, Flato B, Lahdenne P, Michels H, Murray KJ, Punaro L, Rennebohm R, Russo R, Balogh Z, Rooney M, Pachman LM, Wallace C, Hashkes P, Lovell DJ, Giannini EH, Gare BA, Martini A; Paediatric Rheumatology International Trials Organisation (PRINTO); Pediatric Rheumatology Collaborative Study Group (PRCSG). The Paediatric Rheumatology International Trials Organisation provisional criteria for the evaluation of response to therapy in juvenile dermatomyositis. Arthritis Care Res (Hoboken). 2010 Nov;62(11):1533-41. doi: 10.1002/acr.20280. Epub 2010 Jun 25. PMID 20583105
- [Background] Lazarevic D, Pistorio A, Palmisani E, Miettunen P, Ravelli A, Pilkington C, Wulffraat NM, Malattia C, Garay SM, Hofer M, Quartier P, Dolezalova P, Penades IC, Ferriani VP, Ganser G, Kasapcopur O, Melo-Gomes JA, Reed AM, Wierzbowska M, Rider LG, Martini A, Ruperto N; Paediatric Rheumatology International Trials Organisation (PRINTO). The PRINTO criteria for clinically inactive disease in juvenile dermatomyositis. Ann Rheum Dis. 2013 May;72(5):686-93. doi: 10.1136/annrheumdis-2012-201483. Epub 2012 Jun 26. PMID 22736096
- [Derived] Curiel RV, Nguyen W, Mamyrova G, Jones D, Ehrlich A, Brindle KA, Haji-Momenian S, Sheets R, Kim H, Jones OY, Rider LG; Abatacept in Dermatomyositis (AID) Trial Investigators. Improvement in Disease Activity in Refractory Juvenile Dermatomyositis Following Abatacept Therapy. Arthritis Rheumatol. 2023 Jul;75(7):1229-1237. doi: 10.1002/art.42450. Epub 2023 Jun 7. PMID 36657109

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label (One Arm): A patient's participation in this open label non-randomized trial will last approximately 24 weeks (Screening visit and 5 intervention visits) with possible extension to 48 weeks. At screening, participants will have a physical exam, muscle strength assessment, blood and urine collection, and chest x-ray; they will also be asked to complete several questionnaires. All participants will receive each week subcutaneous injection of Abatacept. During intervention phase of the trial, muscle strength testing, physical exam, disease activity measurements, blood and urine collection, and muscle MRI will be performed. Participants will also be asked to complete several questionnaires. Participants will be also monitored closely for for serious drug related side effects.
  Abatacept: Study participation will consist of a screening visit and 5 protocol visits over six months (week 0, week 6, week 12, week 18, and week 24) for each subject, and phone follow-up (week 2, week 4, week 8, week 10, week 14, week 16, week 20, and week 22). At Visit 1, which will be treatment initiation, eligible subjects will be instructed on the use and side effects of subcutaneous abatacept and will be started on the study drug (abatacept 125 mg SQ weekly for subjects with body weight ≥ 50 KG or abatacept 87.5mg SQ for subjects with body weight < 50 KG).
Period: Overall Study
Arm/Group | Open Label (One Arm)
Started | 10
Completed | 9 (One patient did not receive Abatacept at week 24 due to worsening pre-existing ILD.)
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Open Label (One Arm): Subcutaneous abatacept (125 mg weekly for ≥50 kg and 87.5 mg weekly for <50 kg) in combination with standard treatment for 24 weeks (6 months)
Arm/Group | Open Label (One Arm)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 12.0 [7.1 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Meeting the Definition of Improvement (DOI) at Week 24: at Least 3 of 6 Core Set Measures (CSM) Improved by ≥ 20% With no More Than 2 CSM Worsening by ≥ 25% (Not Including the Manual Muscle Testing).
Description: Improvement in myositis disease activity will be assessed using the IMACS myositis definition of improvement (DOI): at least 3 of 6 Core Set Measures (CSM) improved by ≥ 20% with no more than 2 CSM worsening by ≥ 25% (a worsening measure cannot be the manual muscle testing (MMT).
Time Frame: week 0 to week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label (One Arm)
Number analyzed (Participants) | 10
Participants
  Met DOI | 9
  Did not Meet DOI | 1

2. Primary Outcome: Number of Treatment-emergent Adverse Events
Description: Safety will be assessed by review of adverse events using NCI Common Terminology criteria v5.0 November 2017. Particular attention to serious adverse events and infections will be given. An adverse event diary will be maintained throughout the study. Patient evaluations will include: vital sign measurement, physical examination, and laboratory parameters for hematology and routine chemistries
Time Frame: week 0 to week 24
Measure: Number; unit: events
Arm/Group | Open Label (One Arm)
Number analyzed (Participants) | 10
events
  Worsening of interstitial lung disease | 1
  Compression fracture | 1
  Right knee contracture worsening | 1
  Worsening calcinosis | 2
  Lipoatrophy, focal | 1
  Febrile episodes | 2
  Skin-infection | 1
  E. coli diarrhea | 1

3. Secondary Outcome: Total Improvement Score by IMACS Core Set Measures at Week 24
Description: The ACR-EULAR Response Criteria use a continuous total improvement score from baseline (range 0-100) based on the sum of the absolute percent change in the 6 core domains (weighted) used in the IMACS DOI (International Myositis Assessment and Clinical Studies definition of improvement)
  IMACS core measures are: Physician Global Assessment of Disease Activity (PGA), Patient (Subject) Global Assessment of Disease Activity (SGA), Manual Muscle Test (MMT-8), Health Assessment Questionnaire-Disability Index (HAQ-DI), Muscle Enzyme levels, Myositis Disease Activity Assessment Tool (MDAAT) Extramuscular Global Activity.
  In children, the total improvement score ranges between 0 and 100 percent corresponds to the degree of improvement, with higher scores corresponding to a greater degree of improvement ( >/= 30 represents minimal improvement, a score of >/= 45 represents moderate improvement, and a score of >/= 75 represents major improvement).
Time Frame: week 0 to week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label (One Arm)
Number analyzed (Participants) | 10
score on a scale | 53.8 (19.2)

4. Secondary Outcome: Change in Corticosteroid Dose for Steroid-sparing Benefit From Baseline to Week 24
Description: Patients who have achieved Definition of Improvement (DOI) at week 6 (visit 2) or at any point thereafter and is rated by their study physician as at least minimally improved, then tapering of corticosteroids may commence using a precise dose reduction schedule as follows:
  For patients taking 40 to 60 mg daily, prednisone will be tapered by 10 mg ,For patients taking 20 to 35 mg daily, prednisone will be tapered by 5 mg. For patients taking 7.5 to 15 mg daily, prednisone will be tapered by 2.5 mg. For patients taking 1 to 5 mg daily, prednisone will be tapered by 1 mg For patients receiving intravenous pulse methylprednisolone therapy, they may alternatively reduce the dose of IV therapy, instead of oral by a decrease of 25%
Time Frame: week 0 to week 24
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Week 0 (Baseline): Subjects at baseline
- Week 24: Subjects at end of trial
Arm/Group | Week 0 (Baseline) | Week 24
Number analyzed (Participants) | 10 | 10
mg | 16.7 (7.5) | 10.2 (5.4)
Statistical Analysis 1: Comparison: Week 0 (Baseline) vs Week 24; Test type: Other; p = 0.002, t-test, 2 sided

5. Secondary Outcome: Improvement in Physician Global Activity From Baseline to Week 24
Description: This tool measures the global evaluation by the treating physician of the overall disease activity of the patient at the time of assessment using a 10 cm visual analogue scale (VAS). Physician global activity ranges between 0 and 10 via VAS. Lower scores indicate less disease activity.
Time Frame: week 0 to week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Week 0 (Baseline) | Week 24
Number analyzed (Participants) | 10 | 10
units on a scale | 5.0 (1.0) | 2.6 (1.5)
Statistical Analysis 1: Comparison: Week 0 (Baseline) vs Week 24; Test type: Other; p < 0.001, t-test, 2 sided

6. Secondary Outcome: Improvement in Parent/Patient Global Activity From Baseline to Week 24
Description: This tool measures the global evaluation y the patient, or by the parent if the patient is a minor, of the patient's overall disease activity at the time of assessment using a 10 cm. visual analogue scale (VAS). Parent/Patient Global Activity ranges between 0 and 10 via VAS. Lower scores indicate less disease activity.
Time Frame: week 0 to 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Week 0 (Baseline) | Week 24
Number analyzed (Participants) | 10 | 10
units on a scale | 5.3 (1.2) | 2.3 (2.4)
Statistical Analysis 1: Comparison: Week 0 (Baseline) vs Week 24; Test type: Other; p = 0.004, t-test, 2 sided

7. Secondary Outcome: Improvement in Manual Muscle Testing (MMT8) From Baseline to Week 24
Description: Muscle strength will be measured using an abbreviated Manual Muscle Testing (MMT) in 8 muscles (MMT8) ranging between 0 and 10 for each muscle bilaterally (with the exception of neck flexors, for a total of 15 muscles) with a total score ranging between 0 and 150. Higher scores indicate higher muscle strength.
Time Frame: week 0 to week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Week 0 (Baseline) | Week 24
Number analyzed (Participants) | 10 | 10
units on a scale | 121.8 (14.8) | 137.2 (10.7)
Statistical Analysis 1: Comparison: Week 0 (Baseline) vs Week 24; Test type: Other; p < 0.001, t-test, 2 sided

8. Secondary Outcome: Improvement in Childhood Health Assessment Questionnaire (CHAQ) From Baseline to Week 24
Description: Physical function will be measured by using the Stanford HAQ/CHAQ: Childhood Health Assessment Questionnaire: The Stanford HAQ is a brief self-report questionnaire assessing physical function pertaining to activities of daily living in a variety of domains. The CHAQ was adapted directly from the HAQ and it has also been successfully applied to patients with juvenile myositis, with scores ranging from 0 to 3. Lower scores indicate less physical disability.
Time Frame: week 0 to 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Week 0 (Baseline) | Week 24
Number analyzed (Participants) | 10 | 10
units on a scale | 1.84 (0.58) | 0.88 (0.6)
Statistical Analysis 1: Comparison: Week 0 (Baseline) vs Week 24; Test type: Other; p < 0.001, t-test, 2 sided

9. Secondary Outcome: Improvement in Muscle Enzymes From Baseline to Week 24
Description: The muscle enzymes include creatine kinase (CK), aldolase, lactate dehydrogenase (LDH), alanine aminotransferase (ALT) and aspartate aminotransferase (AST). If more than one muscle enzyme is identified as being elevated (a minimum level of 1.3 x the upper limit of normal), then the most abnormal will be selected and this enzyme will be the target enzyme followed to evaluate disease improvement or worsening.
  In order to standardize the change in muscle enzymes selected as most abnormal across patients, the outcome measurement was calculated as the most abnormal enzyme level measured via bloodwork divided by the upper limit normal of the healthy reference range (i.e percentage of the upper limit normal for the respective muscle enzyme). Higher percentages indicate higher muscle enzyme levels.
Time Frame: week 0 to 24
Measure: Mean (Standard Deviation); unit: percentage of upper limit normal
Arm/Group | Week 0 (Baseline) | Week 24
Number analyzed (Participants) | 10 | 10
percentage of upper limit normal | 1.52 (0.66) | 1.52 (1.17)
Statistical Analysis 1: Comparison: Week 0 (Baseline) vs Week 24; Test type: Other; p = 0.375, t-test, 2 sided

10. Secondary Outcome: Improvement in Extramuscular Activity From Baseline to Week 24
Description: The extramuscular activity will be measured by using the Myositis Disease Activity Assessment Tool (MDAAT). This validated tool measures the degree of disease activity of extra-muscular organ systems and muscle on a 0 - 10 cm visual analogue scale (VAS). Extramuscular activity ranges between 0 and 10 via VAS. Lower scores indicate lower disease activity.
Time Frame: week 0 to 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Week 0 (Baseline) | Week 24
Number analyzed (Participants) | 10 | 10
units on a scale | 4.1 (1.5) | 2.4 (1.7)
Statistical Analysis 1: Comparison: Week 0 (Baseline) vs Week 24; Test type: Other; p < 0.001, t-test, 2 sided

11. Secondary Outcome: Improvement in Cutaneous Disease Activity From Baseline to Week 24
Description: Cutaneous disease activity will be measured using the Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI). CDASI is a clinician-scored instrument that separately measures activity and damage in the skin of dermatomyositis patients for use in clinical practice or clinical/therapeutic studies. Cutaneous disease activity was measured via the activity sub-score of CDASI, ranging from 0-100. Higher scores indicate more disease activity.
Time Frame: week 0 to week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Week 0 (Baseline) | Week 24
Number analyzed (Participants) | 10 | 10
score on a scale | 21.4 (11.0) | 14.0 (8.6)
Statistical Analysis 1: Comparison: Week 0 (Baseline) vs Week 24; Test type: Other; p = 0.044, Sign test; Data was not normally distributed

12. Secondary Outcome: Improvement in Total Muscle Edema by MRI From Baseline to Week 24
Description: Axial STIR and T1 MRI images of bilateral thighs and pelvis were obtained at baseline and week 24. Images were coded and reviewed independently by two musculoskeletal radiologists who had comparable inter-observer variability and were blinded to any subject data, including visit number. MRI scoring was performed utilizing a 4-point scale (0-normal, 1-mild, 2-moderate, 3-severe) for muscle edema for each of the muscle groups examined, i.e. gluteal, adductors, hamstrings, and quadriceps, resulting in an aggregate score between 0 to 12.
Time Frame: week 0 to week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Week 0 (Baseline) | Week 24
Number analyzed (Participants) | 10 | 10
score on a scale | 5.3 (3.5) | 2.3 (2.6)
Statistical Analysis 1: Comparison: Week 0 (Baseline) vs Week 24; Test type: Other; p = 0.01, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: week 0 to week 24
Groups:
- Open Label Abatacept: A patient's participation in this open label non-randomized trial will last approximately 24 weeks (Screening visit and 5 intervention visits) with possible extension to 48 weeks. At screening, participants will have a physical exam, muscle strength assessment, blood and urine collection, and chest x-ray; they will also be asked to complete several questionnaires. All participants will receive each week subcutaneous injection of Abatacept. During intervention phase of the trial, muscle strength testing, physical exam, disease activity measurements, blood and urine collection, and muscle MRI will be performed. Participants will also be asked to complete several questionnaires. Participants will be also monitored closely for for serious drug related side effects.
  Abatacept: Study participation will consist of a screening visit and 5 protocol visits over six months (week 0, week 6, week 12, week 18, and week 24) for each subject, and phone follow-up (week 2, week 4, week 8, week 10, week 14, week 16, week 20, and week 22). At Visit 1, which will be treatment initiation, eligible subjects will be instructed on the use and side effects of subcutaneous abatacept and will be started on the study drug (abatacept 125 mg SQ weekly for subjects with body weight ≥ 50 KG or abatacept 87.5mg SQ for subjects with body weight < 50 KG).
Arm/Group | Open Label Abatacept
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Abatacept (N=10)
Worsening of interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Compression fracture (Musculoskeletal and connective tissue disorders) | 1
Calcinosis (Skin and subcutaneous tissue disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Abatacept (N=10)
Right knee contracture worsening (Musculoskeletal and connective tissue disorders) | 1 (1)
Lipoatrophy, focal (Skin and subcutaneous tissue disorders) | 1 (1)
Febrile episodes (General disorders) | 2 (2)
Skin-infection (Skin and subcutaneous tissue disorders) | 1 (1)
E. coli diarrhea (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Non-randomized open label study design

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT02594735/Prot_SAP_000.pdf